CLINICAL TRIAL: NCT01775085
Title: Development of Group Interventions for Breast Cancer Survivors
Brief Title: Group Interventions for Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-291
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Survivor
Keywords: Interventions; Meaning-Centered Group (MCG); Discussion Group (DG); Modules; Sessions; 12-291

ARMS (2):
- Meaning-Centered Group for Breast Cancer Survivors (MCG-BCS) (Experimental)
  Interventions: Behavioral: manualized group intervention
- Discussion Group (DG) (Active Comparator)
  Interventions: Behavioral: standardized, manualized group intervention

INTERVENTIONS:
Behavioral: manualized group intervention — MCG-BCS manual outlines 8 approximately, 90-minute modules: 1) Concepts & Sources of Meaning; 2) Identity, Cancer Survivorship, & Meaning; 3) Historical Sources of Meaning: Past Legacy; 4) Historical Sources of Meaning: Present & Future Legacy; 5) Attitudinal Sources of Meaning: Encountering Life's Limitations; 6) Creative Sources of Meaning: Creativity & Responsibility; 7) Experiential Sources of Meaning: Connecting with Life via Love, Beauty, & Humor; and 8) Transitions: Reflections & Hopes for the Future.
  Arms: Meaning-Centered Group for Breast Cancer Survivors (MCG-BCS)
Behavioral: standardized, manualized group intervention — DG is a standardized, manualized group developed by the MSKCC Psychiatry Service and utilized in a similar form in our completed and ongoing RCTs of MCGP. Based on models described by Rogers and Bloch, the essential components include reassurance, explanation, education, encouragement, and permission for expression. The process emphasizes Rogerian concepts (e.g., empathic understanding) and avoids techniques that are not exclusively supportive. The content focuses on education about here-and-now topics relevant to BCS (e.g., maintaining and eliciting social support, financial strains, return to work, physical symptom management), allowing emotional expression and discussion of difficult topics.
  Arms: Discussion Group (DG)

SUMMARY:
The purpose of this study is to compare two types of groups for breast cancer survivors: a Meaning-Centered Group and a Discussion Group. Many breast cancer survivors seek help to deal with the emotional burden of having gone through the cancer experience. Participation in groups offering support often helps cancer survivors cope with stressors of life after having had cancer by giving them a place to express their feelings. The "Meaning-Centered Group" is intended to teach breast cancer survivors how to maintain or even increase a sense of meaning and purpose in their lives after treatment for cancer. The "Discussion Group" is intended to help breast cancer survivors cope by giving them a place to get support from other breast cancer survivors.

The goal of this study is to compare the benefits of these two types of group approaches for breast cancer survivors. The study is also testing the benefits and feasibility of conducting the groups virtually using a telephone and computer.

ELIGIBILITY:
Inclusion Criteria:

* History of non-metastatic breast cancer (DCIS or Stage I, II, or III) as recorded in the medical record at MSKCC by self-report, or by outside correspondence, including a study checklist signed by a physician for patients outside of MSKCC
* Post completion of treatment (may be on hormone therapy, such as Tamoxifen or monoclonal antibody, such as Herceptin or Pertuzumab)) for any type of cancer as confirmed by the medical record at MSKCC, by self-report, or by outside correspondence, including a study checklist signed by a physician for patients outside of MSKCC
* Age 18 or older
* Access to a telephone, computer (e.g. desktop, laptop, smartphone, tablet) and Internet

For Phase 2 only:

* A score of ≥ to 4 on the Distress Thermometer (DT) and indication that this distress is related in some way to the patient's breast cancer or survivorship
* If taking medication for mood, anxiety, depression, thoughts, sensory experiences such as hallucinations, or sleep, stable and consistent enough in dosage and use of that medication so as to not result in a clinically significant change as determined by the study PI/co-PI or, confirmed by reports in the medical record at MSKCC, by selfreport, or by outside correspondence, including a study checklist signed by a physician for patients outside of MSKCC
* Did not participate in Phase 1

Exclusion Criteria:

* Evidence of or treatment metastatic disease
* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent or participating in the groups (i.e., acute psychiatric symptoms which require individual treatment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
feasibility as measured by the proportion of patients enrolled who complete 4 out of 8 modules, which should not be not lower than 40%. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Monique James, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/